CLINICAL TRIAL: NCT07198958
Title: Immune Adverse Events Registry in Onco-Hematologic Patients Treated With Immunotherapy
Acronym: MITOX
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Roberto Ferrara, Dr. Roberto Ferrara, IRCCS San Raffaele
Other Study IDs: MITOX
Record Dates: First submitted 2025-09-15; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Cancer; Cancer (Colon Cancer, Breast Cancer, Lymphoma, Chronic Lymphoma Leukemia, Multiple Myeloma); Cancer (Solid Tumors); Cancer (With or Without Metastasis)
Keywords: Immunotherapy; Adverse Events; Cancer; Immune-Related Adverse Events; irAEs; PD-1/PD-L1 inhibitors; anti-CTLA-4 agents; ICI
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Breast Neoplasms; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immunotherapy is a therapeutic strategy aimed at inducing the immune system to identify and combat cancer cells and, alongside the evident clinical success observed in many patients, a specific toxicity profile has emerged, associated with the modulation of the immune system achieved with this type of drugs, known as Immune-Related Adverse Events (irAEs). irAEs encompass a highly heterogeneous spectrum of autoimmune manifestations that can potentially involve any organ or system, occurring in ~ 80% of patients treated with anti-CTLA-4 agents and in ~ 60-70% of patients treated with PD-1/PD-L1 inhibitors. However, severe (grade 3-4) irAEs affect only ~ 15% of patients treated with CTLA-4 inhibitors and ~ 5-10% of patients receiving anti-PD-1/PD-L1 agents, with a mortality rate ranging from 0.36% to 1.23%. The main characteristic of irAEs is their unpredictability in terms of time of onset, severity and responsiveness to immunosuppressive agents. Therefore, the management of irAEs often requires clever interpretation of clinical symptoms, proper choice of laboratory tests and imaging tools, and ability to perform differential diagnosis with other condition associated to tumour itself or to unrelated concomitant events (i.e., infections). Although international societies (i.e.; ESMO) have provided detailed guidelines for the management of irAEs or algorithms for the administration of ICI in patients with pre-existing autoimmune disease, they are sometimes difficult to be applied to certain complex situations. Furthermore, given the scarcity of data from clinical trials, some of these recommendations are mainly based on highly heterogeneous patients' population included in relatively small real world studies. Therefore, recommendations should always be adapted to specific clinical conditions and challenges. Studies investigating these aspects have particularly focused on the autoimmune antibody response, correlating its positivity in various ways with clinical outcomes. However, the results across different studies are not consistent. Moreover, additional prospective data are needed to confirm which information can guide the management of irAEs in order to optimize therapy and improve prognosis without negatively impacting oncological outcomes. The adoption of a therapeutic strategy tailored to irAEs is essential for improving both the immunological and oncological prognosis of patients affected by this group of manifestations. A prospective and cross-sectional observational approach to study irAEs is fundamental to the development of such therapeutic innovation. This study approach must be based not only on monitoring patients who have already developed irAEs but also on profiling patients even before the development of irAEs to determine which factors are associated with this group of pathologies and the different characteristics they may assume once they arise. The protocol will be based on the retrospective acquisition of data concerning the clinical history of the patients involved, from birth until recruitment into the study, and the prospective recording of information regarding the disease characteristics (both immuno-rheumatological and oncological) and the subsequent evolution of the clinical picture. Study procedures will take place during visits scheduled as part of routine clinical practice and will include the collection of data-clinical, laboratory, and imaging-related to the patient's oncological disease and irAEs, the characteristics of the diagnostic-therapeutic procedures performed, and the subsequent immuno-oncological outcomes. All patients scheduled to begin immunotherapy treatment will be enrolled in the study, as well as those who have developed irAEs without being enrolled prior to the onset of immuno-mediated manifestations. Enrolled patients who do not develop irAEs will be considered as the control group, providing essential information on risk profiling for the development of irAEs.

DETAILED DESCRIPTION:
Immunotherapy is a therapeutic strategy aimed at inducing the immune system to identify and combat cancer cells. The rationale behind immunotherapy lies in the context of an altered homeostasis between the immune system and cancer, where the latter prevails. The goal of this type of therapy is to initiate or restore a cycle in which immunity against the tumor is maintained and can be amplified and propagated to achieve good control over the disease. Immune Checkpoint Inhibitors (ICIs) are monoclonal antibodies used in cancer therapy designed to remove the inhibitory brake imposed on T cells, thereby allowing a robust activation of the immune system against the tumor. Over time, the use of ICIs has become increasingly widespread, and alongside the evident clinical success observed in many patients, a specific toxicity profile has emerged, associated with the modulation of the immune system achieved with this type of drugs, known as Immune-Related Adverse Events (irAEs). irAEs encompass a highly heterogeneous spectrum of autoimmune manifestations that can potentially involve any organ or system. By releasing the brakes on checkpoint controls, monoclonal antibodies targeting CTLA-4 (Cytotoxic T Lymphocyte Antigen - 4) and the PD-1 (Programmed cell Death Protein 1) / PD-L1 (Programmed Death-Ligand 1) axis can activate pre-existing autoreactive T-cells or generate novel autoreactive T-cell clones, triggering immune-related adverse events (irAEs) of various types and severity. IrAEs are common occurring in ~ 80% of patients treated with anti-CTLA-4 agents and in ~ 60-70% of patients treated with PD-1/PD-L1 inhibitors. However, severe (grade 3-4) irAEs affect only ~ 15% of patients treated with CTLA-4 inhibitors and ~ 5-10% of patients receiving anti-PD-1/PD-L1 agents, with a mortality rate ranging from 0.36% to 1.23%. The most common irAEs are those affecting the skin, gastrointestinal tract, and endocrine glands. From a rheumatological perspective, inflammatory arthritis and polymyalgia-like syndromes are the most prevalent forms, while the more severe cases include myositis, which may also involve myocardial complications. The main characteristic of irAEs is their unpredictability in terms of time of onset, severity and responsiveness to immunosuppressive agents . Therefore, the management of irAEs often requires clever interpretation of clinical symptoms, proper choice of laboratory tests and imaging tools, and ability to perform differential diagnosis with other condition associated to tumour itself or to unrelated concomitant events (i.e., infections). Although international societies (i.e.; ESMO) have provided detailed guidelines for the management of irAEs or algorithms for the administration of ICI in patients with pre-existing autoimmune disease , they are sometimes difficult to be applied to certain complex situations. Furthermore, given the scarcity of data from clinical trials, some of these recommendations are mainly based on highly heterogeneous patients' population included in relatively small real word studies. Therefore, recommendations should always be adapted to specific clinical conditions and challenges. As an example, although most of the current international guidelines recommend steroid treatment and permanent discontinuation of ICI after a grade 3 irAEs, retrospective studies have reporting spontaneous resolution of grade 3 immune related hepatitis in up to 50% of patients who temporary withhold ICI without receiving any immunosuppressive treatment . A similar "grey area" in the management of irAEs deals with the impact of steroid sparing strategies such as disease-modifying antirheumatic drugs (DMARDs) on the oncological outcome of cancer patients experiencing irAEs. In fact, while some studies suggested a potential detrimental effect of DMARDs on response with ICI in patients with melanoma and irAEs, the investigators and other groups have reported that tailoring immunosuppression using DMARD in steroid-refractory patients is associated with a good remission rate of irAEs and no negative impact on the oncological outcomes. In addition, the investigators have identified a panel of autoantibodies able to predict the emergency of steroid refractory irAEs, which could help to better select patients for whom an earlier upfront tailored management of irAEs could be required.

Despite recommendations from major European and American rheumatology and oncology societies regarding the management of irAEs, these guidelines are largely based on expert opinion, and this complex group of manifestations remains challenging to treat. In recent years, potential predictors have been identified, both in terms of the likelihood of developing irAEs and concerning clinical characteristics and responses to available therapies. Studies investigating these aspects have particularly focused on the autoimmune antibody response, correlating its positivity in various ways with clinical outcomes. However, the results across different studies are not consistent. Additionally, both prospective and retrospective studies have led to very different conclusions, and these predictive factors have not yet been implemented in clinical practice . As a result, the therapeutic algorithm in this clinical scenario remains highly variable and often unsatisfactory. Furthermore, it has not yet been conclusively determined whether immunosuppressive therapies administered to patients with irAEs have a negative impact on oncological prognosis. In this regard, there is also a lack of data on the role of continuing immunotherapy in patients with irAEs and whether this strategy could mitigate the aforementioned impact.

A multidisciplinary case-by-case approach involving oncologist and organ-specialists is likely to lead to an optimal tailored decision for each patient. Several published experiences from the Gustave Roussy Cancer Campus, the Johns Hopkins University School of Medicine and the Belgian Society of Medical Oncology have reported that multidisciplinary managements of irAEs are feasible, could facilitate a prompt resolution of irAEs and could generate knowledge in the field (i.e.; ~ 6% of irAEs discussed at multidisciplinary level were classified as novel and unexpected events). In this regard, multidisciplinary management of irAEs could constitute a forum with a high educational value deriving from a cross-fertilization between different fields of medicine. As an example, attendance by organ specialists could provide them new insights into the pathophysiological features of autoimmune diseases in non-cancer patients Therefore, additional prospective data are needed to confirm which information can guide the management of irAEs in order to optimize therapy and improve prognosis without negatively impacting oncological outcomes. The adoption of a therapeutic strategy tailored to irAEs is essential for improving both the immunological and oncological prognosis of patients affected by this group of manifestations. A prospective and cross-sectional observational approach to studying irAEs is fundamental to the development of such therapeutic innovation. This study approach must be based not only on monitoring patients who have already developed irAEs but also on profiling patients even before the development of irAEs to determine which factors are associated with this group of pathologies and the different characteristics they may assume once they arise. However, this study approach requires the integration of multiple clinical competencies to cover the extensive clinical-pathological spectrum that characterizes irAEs, as well as the complexity of concomitant neoplastic diseases and oncological pharmacology.

Such a process is potentially easier to implement in clinical settings like the Units of Immunology, Rheumatology, Allergy and Rare Diseases (UniRAR), Oncology, Urology, and Gynecology at San Raffaele Hospital, where the concurrent presence of expertise in both immuno-rheumatology and oncology-supported by constant interdisciplinary dialogue-is a structural reality.

The results generated by this complex experimental strategy could lead to a redefinition of the current diagnostic and therapeutic paradigm for irAEs.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female patient (≥18 years old) with diagnosis of solid or hematologic tumor scheduled to begin immunotherapy treatment (prospective)
* Any male or female patient (≥18 years old) with diagnosis of solid or hematologic tumor already in treatment with immunotherapy with development of irAEs (retro/prospective)
* Any male or female patient (≥18 years old) with diagnosis of solid or hematologic neoplasm previously treated with immunotherapy and history of irAEs (retrospective)
* Patients able to understand and sing an informed consent form (prospective group)

Exclusion Criteria:

* Patients < 18 years of age
* Patients with uncertain diagnosis of solid or hematologic tumor
* Patients not eligible for any clinical reason for immunotherapy
* Patients unable to understand or sign an informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of all ages, 18 years and older, with diagnosis of solid or hematologic tumor scheduled to begin immunotherapy treatment or with development of irAEs while treated with immunotherapy.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2045-09 (Estimated); Study Completion 2045-09 (Estimated)

PRIMARY OUTCOMES:
Incidence and characterization of irAEs, from diagnosis to treatment | Data will be collected at baseline, at the onset of irAEs, and at their resolution. Survival and response to oncological treatment will be updated throughout patient follow-up until study completion, with the registry planned to run for 20 years.
  The registry aims to characterize the phenotype of patients for the diagnosis and treatment of irAEs by collecting a wide range of data-clinical, laboratory (including tissue samples, PBMCs, plasma, serum, and autoantibody profiles), and imaging-regarding predictive factors, presenting manifestations, and the evolution of adverse events according to the type and and grade of irAE (measured according to CTCAE v5.0). Data will also include diagnostic-therapeutic strategies adopted, such as type and dosage of immunosuppressive therapy, autoimmune markers tested, and imaging parameters, as well as oncological outcomes such as OS, PFS (measured in months) and ORR (measured as the percentage of patients achieving complete or partial response according to RECIST v1.1). This comprehensive data collection will allow subsequent correlations between baseline characteristics, treatment strategies, and both immunological and oncological outcomes.

SECONDARY OUTCOMES:
Assessing the effectiveness of irAE management | Data will be collected at baseline, at the onset of irAEs, and at their resolution. Survival and response to oncological treatment will be updated throughout patient follow-up until study completion, with the registry planned to run for 20 years.
  Furthermore, the registry will aim to evaluate the effectiveness of diagnostic and therapeutic multidisciplinary management currently considered the gold standard in clinical practice for irAEs, comparing these real-world practices with published guideline-based approaches by assessing clinical resolution rates of irAEs (percentage of resolved events). It will also seek to identify potential areas for improvement in these practices for the overall patient population or for specific patient subgroups defined by baseline characteristics, to better understand variability in management outcomes. In addition, the registry will correlate the aforementioned information to enhance knowledge of the pathophysiology of irAEs, including the role of predictive biomarkers and immunological signatures, and will assess the impact of different irAE management strategies on oncological outcomes such as response to immunotherapy, thus clarifying whether tailored immunosuppressive approaches